CLINICAL TRIAL: NCT02909543
Title: The Life Experience of Young Women (Age 18-38) Who Live With Congenital Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 51-2016
Record Dates: First submitted 2016-09-01; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-05

CONDITIONS: Women With Congenital Heart Diseases
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Other: Observation and Interviwe — The research data will be conducted by using a semi structured interview of the participants in the study.

SUMMARY:
This research will focus on young women between the ages of 18-38 who underwent a heart operation and their life experiences. This research will focus on these life events and the paradigm of these women being raised as "heart sick," and consequently lacking self-esteem (Frigiola, Bull, & Wray, 2014; Hickey et al., 2012). Most qualitative studies focusing on the quality of life compare men and women, completely ignoring women's body image and the experience of womanhood (Hickey et al., 2012; Hövels-Gürich et al., 2007; Sarikouch, et al., 2013). This study aims to focus on women's stories about their life experiences and the influence of surgery(ies) on their daily life using an the qualitative phenomenological approach.

ELIGIBILITY:
Inclusion Criteria:

* Atrial septal defect or ASD,
* Ventricle septal defect or VSD,
* Tetralogy of Fallot or TOF
* Translocation of great arteries or TGA
* underwent heart operation
* Hebrew speakers that are able to understand the meanings of the questions and tell their life stories.

Exclusion Criteria:

* Non Hebrew speakers
* Did not underwent heart surgery.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study aims to focus on women's stories about their life experiences and the influence of surgery(ies) on their daily life using an the qualitative phenomenological approach.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Interview about the life experience of young women (age 18-38) who live with congenital heart disease and overwent an open heart operation. | 1day, at the time of the interview

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe MC,, Hadera, Israel